CLINICAL TRIAL: NCT04970017
Title: Correlation Between Left Ventricular Global Strain Measured by Speckle Tracking Echocardiography and Scar Burden Measured by Cardiac Magnetic Resonance Imaging in Patients With Ischemic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Mohamed Abdellatif, Dr, Assiut University
Other Study IDs: 17200538
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-02

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Cardiac MRI, Echocardiography — Magnetic resonance imaging, Echocardiography

SUMMARY:
To verify whether GLS and LV mechanical dispersion, measured by two-dimensional speckle-tracking echocardiography (2D-STE) correlate with LV scar burden measured by cardiac MRI in patients with ischemic heart disease.

DETAILED DESCRIPTION:
Evaluation of presence, localization, and extent of left ventricular(LV) scar tissue in patients with ischaemic heart disease (IHD) is of fundamental importance in clinical practice. It affects the decision making regarding revascularization and is a determinant of subsequent mortality. (Mele, Fiorencis et al. 2016) Late gadolinium contrast-enhanced cardiac magnetic resonance (LGE-CMR) is considered the current gold standard technique for assessment of the scar burden in IHD patients. However, it is not readily accessible in many areas due to availability and cost issues.(Abou, Prihadi et al. 2020), (Bendary, Afifi et al. 2019) Several recent studies suggested 2-D speckle tracking strain as a potential surrogate for cardiovascular magnetic resonance (CMR) late gadolinium enhancement (LGE) imaging. This would be useful in cases where CMR is not available, gadolinium contrast is contraindicated, or in patients at greater risk of adverse long term events. (Erley, Genovese et al. 2019) Among echocardiography derived strain measurements, global longitudinal strain (GLS) was shown to be superior to global circumferential strain (GCS) in its ability to detect subtle myocardial abnormalities due to better reproducibility (Erley et al, 2019). Left ventricular mechanical dispersion (LVMD) is also considered a valuable parameter that was associated with outcomes after myocardial infarction. (Abou, Prihadi et al. 2020).

Despite the growing number of strain related studies in the literature, it is not clear whether the relationship of strain measurements with LGE is strong enough for strain to be considered as a surrogate. (Erley, Genovese et al. 2019). Also, the differences between GLS and LV MD among strain components in this context are not well established.

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting for viability assessment in to cardiac MRI unit, Assiut university heart hospital, with a history of previous stemi, at least 3 months after the acute event ( scar stabilization) and up to one year

Exclusion Criteria:

* Patients with:

  * Contraindication to cardiac MRI (claustrophobia, Patients with eGFR below 30 mL/min/1.73 m2. and patients with metallic implants)
  * Non-ischemic cardiomyopathy.
  * Valvular heart disease (VHD).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting for viability assessment in to cardiac MRI unit, Assiut university heart hospital, with a history of previous stemi, at least 3 months after the acute event ( scar stabilization) and up to one year
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Scare burden by echocardiography | One year
  To test the correlation between the scar burden measured by cardiac MRI and GLS measured by 2D STE

SECONDARY OUTCOMES:
Value of spickle tracking echocardiography in clinical practice | One year
  Predicting the scar burden in ICMP patients by GLS and mechanical dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdellatif, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt